CLINICAL TRIAL: NCT04808908
Title: Effect of N-803 on B Cell Follicles in Antiretroviral Treated HIV Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDIM-2019-27395; 5UM1AI126611 (NIH)
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Hiv; HIV Infections; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N-803 (Experimental): All participants will receive the intervention, N-803 treatment.
  Interventions: Biological: N-803

INTERVENTIONS:
Biological: N-803 — N-803, provided by ImmunityBio., Inc. will be administered subcutaneously at a dose 6 mcg/kg on Days 0, 21, and 42 (with a dosing window of up to 14 days post the planned dosing day)

SUMMARY:
N-803 has demonstrated ability to reactivate HIV from latency and can activate T cells and NK cells to clear those cells, thus reducing the reservoir. However, a concern is that CD8 T cells may be excluded from the B cell follicles, where a significant part of the reservoir resides. Webb, et al, has shown that in SIV infected monkeys CD8 T cells in follicles increase in frequency when N-803 is administered. We hypothesize that in HIV infected humans treated with N-803 that CD8 T cells will increase in B cell follicles and that there will be a further reduction in the frequency of cells with an inducible provirus.

DETAILED DESCRIPTION:
A phase 1B single arm study of 10 HIV-infected adults on effective ART will be performed. This is a two-center, non-randomized, open label, and uncontrolled study.

All participants will undergo an extensive baseline evaluation 7-14 days before the first dose that will include an excisional biopsy of a lymph node, colonic biopsies, and leukapheresis. Participants will then receive three doses of N-803 administered every 21 days. A second excisional biopsy will be performed between 7-14 days after the final dose. The study drug N-803 will be administered at 6 mcg/kg, which is the maximum tolerated dose determined in a recently completed dose-escalation study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load.
* On continuous antiretroviral therapy for over 24 months without any interruptions of greater than 14 consecutive days, without plans to modify ARTduring the study period.
* Screening plasma HIV RNA levels < 20 copies/mL and on at least 1 determination in past 12 months (isolated single values greater than or equal to 20 but < 200 copies/mL will be allowed if they were preceded and followed by undetectable viral load determinations)
* Screening CD4+ T cell count greater than or equal to 350 cells/mm3 and nadir CD4+ T cell count of >200 per participant report.
* Ability to be off prednisone and other immunosuppressive drugs for at least 14 days before screen. Inhaled, nasal spray, and topical steroids are acceptable.
* Acceptable blood pressure and heart rate parameters within normal limits (systolic = 88-140mmHg; diastolic = 50-<90mmHg; heart rate = 46-100 bpm). Treatment with antihypertensive medication is allowed. However, if someone is on a beta-blocker this must be switched to another class of medication as there is a theoretical risk for bradycardia if the participant were to experience cytokine release syndrome symptoms (which has not happened with this drug delivered SQ).
* Sexually active females of child bearing potential and males with partners of child bearing potential must agree to use effective contraception during study participation and for 1 month following the final study visit (4 months after final dose of study drug). Acceptable birth control is defined as the following:

  (1) For female participants of childbearing potential, two of the following forms of contraception are required, one of which must be a barrier method:
  1. Condoms (male or female) with or without a spermicidal agent
  2. Diaphragm or cervical cap with spermicide
  3. Intrauterine device (IUD) with published data showing that expected failure rate is < 1% per year
  4. Tubal ligation
  5. Hormone-based contraceptive such as oral birth control pills
* Laboratory tests performed within 14 days of study enrollment must be a grade 0 or 1 as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, with the following exceptions:

  1. Platelet counts (≥ 150,000/mm3)
  2. Hemoglobin > 12.5 g/dL for men and > 11.5 g/dL for women. It is not acceptable for patients to be transfused to meet this requirement. The use of Epogen is permitted.
  3. Estimated Cr Cl (eGFR) > 50

Exclusion Criteria:

* Active or recent malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months; minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) are not exclusionary
* Chronic liver disease defined as Class B and C on the Child-Pugh chronic liver disease scale.
* Active and poorly controlled atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 ACC/AHA guidelines, including a previous diagnosis of any of the following:

  1. acute myocardial infarction
  2. acute coronary syndromes
  3. stable or unstable angina
  4. coronary or other arterial revascularization
  5. stroke
  6. transient ischemic attack (TIA)
  7. peripheral arterial disease presumed to be of atherosclerotic origin.
* History of potential immune-mediated medical conditions requiring concomitant treatment with immunomodulatory drugs, and/or exposure to any immunomodulatory drug in the 30 days prior to screen (e.g. corticosteroid therapy equal to or exceeding a dose of 15 mg/day of prednisone for more than 10 days, IL-2, interferon, methotrexate, cancer chemotherapy). NOTE: use of inhaled, nasal steroid or topical steroid lotions and creams is not exclusionary. Prior exposure to N-803 is not exclusionary if prior exposure occurred at least 6 months before screen.
* Unable to undergo leukapheresis procedure
* Exposure to any experimental therapies within 90 days of study screen. Exposure to long acting injectable ART therapies is not exclusionary.
* Latent TB infection or active TB disease prior to completing a standard regimen of anti-TB therapy that is defined as meeting PPD criteria for TB exposure or a positive quantiferon gold test collected at screening.
* Active fungal infection requiring systemic antifungal therapy
* Active herpes outbreak or varicella-zoster virus infection requiring episodic treatment
* Chronic active hepatitis B or C. For Hepatitis B this will be defined as HBs antigen + and for Hepatitis C this will be defined as Hepatitis C antibody positive and Hepatitis C PCR+.
* History and/or presence of any clinically significant disease or disorder, such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal and psychiatric/mental disease/disorder, which, in the opinion of the site Principle Investigator may either put the subject at risk because of participation in the study, influence the results of the study or the subject's ability to participate in the study.
* Any degree of baseline QT/QTc interval prolongation (QTc interval > 450 msec in males and > 470 msec in females.)
* Any ischemic changes seen in the stress treadmill test administered per the discretion of the PI in order to assess any other EKG abnormalities outlined in study protocol
* History or evidence of uncontrollable CNS disease such as dementia, demyelinating disease, Parkinson's, or a CNS degenerative disease that, in the opinion of the site Principle Investigator, may either put the subject at risk because of participation in the study, influence the results of the study or the subject's ability to participate in the study.
* Prior organ allograft or allogeneic transplantation
* Planning or current pregnancy or breastfeeding
* Any clinically indicated vaccination (other than influenza) administered within 14 days of screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Rhein J, Chipman JG, Beilman GJ, Cromarty R, Escandon K, Anderson J, Wieking G, Reichel J, Batres R, Khoruts A, Basting CM, Hinderlie P, Davis ZB, Eaton A, Vaughn BP, Eilkhani E, Safrit JT, Soon-Shiong P, Baker JV, Klatt NR, Deeks SG, Miller JS, Schacker TW. Impact of the IL-15 superagonist N-803 on lymphatic reservoirs of HIV. JCI Insight. 2025 Jun 3;10(13):e190831. doi: 10.1172/jci.insight.190831. eCollection 2025 Jul 8. PMID 40471871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-803
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | N-803
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety (Adverse Event Rate)
Description: Safety is a primary outcome of this phase 1b trial. Safety will be reported as the number of adverse events per participant.
  This includes all adverse events (total regardless of severity)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: adverse events per participant
Arm/Group | N-803
Number analyzed (Participants) | 10
adverse events per participant | 20 (6.2)

2. Secondary Outcome: Frequency of CD8+ T Cells in Follicles
Description: Frequency of CD8+ T cells in B cell follicles will be determined using flow cytometry and reported in units of cells/g tissue
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cells per gram of LN tissue
Arm/Group | N-803
Number analyzed (Participants) | 10
cells per gram of LN tissue | 29400 (26900)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | N-803
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-803 (N=10)
Injection site erythema (General disorders) | 10 (30)
Injection site induration (General disorders) | 4 (6)
Myalgia (General disorders) | 9 (14)
Fatigue or malaise (General disorders) | 8 (13)
Headache (General disorders) | 8 (16)
pain (General disorders) | 7 (10)
lymphadenopathy (Blood and lymphatic system disorders) | 6 (13)
fever (General disorders) | 5 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT04808908/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT04808908/ICF_001.pdf